CLINICAL TRIAL: NCT01361776
Title: Humoral Response to TBE Vaccine in Elderly (50+ Year Olds) After Changed Dosage Intervals/Number of Doses?
Brief Title: Humoral Response to Tick-borne Encephalitis Vaccine in Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Lars Rombo, professor, Sormland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/4-31/2
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Tick-borne Encephalitis
Keywords: immune response; TBE-vaccine; elderly; additional doses
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TBE vaccine at 0+30 days (Active Comparator): This group of 50 participants will follow the standard recommendation and will be given TBE vaccine 0.5 ml FSME immune at 0 + 30 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- TBE vaccine at 0+7+21 days (Active Comparator): This group of 50 participants will will be given TBE vaccine 0.5 ml FSME immune at 0 + 7 +21 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- TBE vaccinte at 0+30+90 days (Active Comparator): This group of 50 participants will will be given TBE vaccine 0.5 ml FSME immune at 0 + 30 + 90 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- younger participants (Active Comparator): This group of 50 participants in the age group 18-49 years will be given TBE vaccine 0.5 ml FSME immune at 0 +30 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune

INTERVENTIONS:
Biological: FSME-immune — 0.5 ml im as scheduled in the 4 arms

SUMMARY:
Antibody titers after tick-borne encephalitis (TBE) vaccination are less in elderly and vaccination breakthroughs are more common in this age group. This has prompted Swedish authorities to recommend an additional dose in the initial vaccination schedule (= 0+30+90 days instead of the usually recommended 0+30 days. The investigators intend to evaluate this regime.

DETAILED DESCRIPTION:
The risk for TBE increases in Sweden. Together with an increased awareness of the possibility to acquire protection by vaccination, this has led to an increase in the number of doses of the vaccine distributed in Sweden each year -now being approximately 400.000. The first year, two doses with an interval of 1 month is recommended for the general population, followed by a third dose approximately one year later and an additional booster dose three years after the third.

Recent studies show that the antibody titers against TBE are substantially less in an older population. This is in line with the present recommendation from Austria that booster intervals should be shortened to 3 years in the age group 60+. It is also in line with a report of vaccination failures where 13/27 patients were older than 60 years According to a study by Jilkowa et al, 18 % (38/185) in the age group 60+ did not achieve putative levels of antibody titers after the first two doses. Therefore, the manufacturer of Encepur recommends a total of three doses to this age group using the same regimen as with "accelerated vaccination schedule (0+7+21 days). Unfortunately, GMT (geometrical mean of titers) after 3 doses with the accelerated schedule are not superior to 2 doses given at 0+30 days.

The manufacturer of FSME-immun instead recommends that serology should be checked one month after the second dose and that a third dose should be given if titers are not sufficient (0+30+60 days). Unfortunately, determinations of titers in a large number of samples put severe strain on logistics and is not feasible in Sweden.

In order to try to improve immunity in the age group 60+ , the Department of Communicable Disease Control and Prevention in Stockholm therefore recommends a third dose two months after the first two doses to the age group 60+ (0+30+60 days).

Study design. The investigators intend to give FSME-immune to 3 groups with varying vaccination schedules ( 0+7+21, 0+30 or 0+30+90. 50 participants will be randomized to each group. Half of them will be between 50-59 years and half will be at least 60 years old. A younger age group (50 participants between 18-49 years) will serve as controls and will be given FSME-immune according to standard recommendations (0+30 days).

Serum samples (10 ml of blood) will be obtained at five times: 0,60,120,360 and 400 days after first dose Samples will be analysed for neutralising antibodies at the Swedish institute for Infectious disease control - other options possible.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or more
* generally healthy
* no immunosuppressive condition
* fertile women must use contraceptives

Exclusion Criteria:

* Previous TBE infection
* Previously immunized with TBE vaccine
* Anaphylactic reaction to egg protein
* Any disease or therapy which might suppress the immune response
* Vaccination should be delayed if a participant has fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Serum concentration of neutralising antibodies against TBE one month after two or three doses. | 18 months after the first dose
  Determination of neutralising antibodies one month after completion of the first years vaccination series

SECONDARY OUTCOMES:
Serum concentration of neutralising antibodies against TBE one month after the dose which will be given a year later | 18 months after the first dose has been given
  Determination of neutralising antibodies one month after the dose which will be given a year later

CONTACTS AND LOCATIONS:
Overall Officials: lars rombo, MD, Principal Investigator — Karolinska Institutet
Locations (6):
- Dept infectious diseases, Helsingfors, Finland
- Sweden (5):
  - Dept infectious diseases, Eskilstuna
  - Dept infectious diseases, Karlstad
  - Department of infectious diseases, Örebro
  - Department of infectious diseases, Stockholm
  - Dept infectious diseases, Uppsala

REFERENCES:
- [Derived] Kantele A, Rombo L, Vene S, Kundi M, Lindquist L, Erra EO. Three-dose versus four-dose primary schedules for tick-borne encephalitis (TBE) vaccine FSME-immun for those aged 50 years or older: A single-centre, open-label, randomized controlled trial. Vaccine. 2022 Feb 23;40(9):1299-1305. doi: 10.1016/j.vaccine.2022.01.022. Epub 2022 Jan 31. PMID 35101266